CLINICAL TRIAL: NCT00976456
Title: Open-label Study of Bevacizumab (Avastin®) in Combination With Pemetrexed or Pemetrexed and Carboplatin as First-line Treatment of Patients With Advanced or Recurrent Non-squamous Non-small Cell Lung Cancer
Brief Title: Efficacy Study of Avastin® With Pemetrexed +/- Carboplatin to Treat Elderly Patients With Non-small Cell Lung Cancer
Acronym: 65plus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PD Dr. med. Wolfgang Schuette (Other)
Collaborators: Roche Pharma AG (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, PD Dr. med. Wolfgang Schuette, PhD MD, Martha-Maria Krankenhaus Halle-Dölau gGmbH
Organization: Martha-Maria Krankenhaus Halle-Dölau gGmbH (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 65 plus; ML21896
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
Keywords: lung cancer; NSCLC; elderly; non-squamous; Elderly patients at least 65 years old; first line therapy; non-squamous non-small cell lung cancer stage IIIb or IV
MeSH Terms: conditions — Lung Neoplasms | interventions — Bevacizumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab + Pemetrexed (Active Comparator): Bevacizumab + Pemetrexed
  Interventions: Drug: Bevacizumab + Pemetrexed
- Bevacizumab + Pemetrexed + Carboplatin (Active Comparator): Bevacizumab + Pemetrexed + Carboplatin
  Interventions: Drug: Bevacizumab + Pemetrexed + Carboplatin

INTERVENTIONS:
Drug: Bevacizumab + Pemetrexed — Bevacizumab 7,5 mg/kg i.v. over 60 min every 3 weeks plus pemetrexed 500 mg/m2 i.v. on D1 over 10 minutes every 3 weeks
  Other Names: Avastin®; ALIMTA®
  Arms: Bevacizumab + Pemetrexed
Drug: Bevacizumab + Pemetrexed + Carboplatin — Bevacizumab 7,5 mg/kg i.v. over 60 min every 3 weeks plus pemetrexed 500 mg/m2 i.v. on D1 over 10 minutes and carboplatin AUC 5 on D1 every 3 weeks
  Other Names: Avastin®; ALIMTA®; Carboplatin
  Arms: Bevacizumab + Pemetrexed + Carboplatin

SUMMARY:
Multi-center, open, randomized (parallel) and comparative phase III.

Eligible patients will receive bevacizumab + chemotherapy for a minimum of 4 cycles followed by bevacizumab (+ pemetrexed, if appropriate) maintenance therapy until disease progression.

Arm A: Bevacizumab + pemetrexed

Arm B: Bevacizumab + pemetrexed + carboplatin

DETAILED DESCRIPTION:
Primary:

* Proof of non-inferior efficacy of a monochemotherapy regimen of pemetrexed plus bevacizumab versus a combination chemotherapy regimen of pemetrexed-carboplatin plus bevacizumab in elderly patients(> 65 years) as first-line treatment of advanced metastatic or recurrent non-squamous NSCLC by progression free survival

Secondary:

* To assess the efficacy of bevacizumab as measured by overall response rate and overall survival.
* To assess the safety of bevacizumab in combination with pemetrexed and pemetrexed and carboplatin.
* To assess quality of life by EORTC questionnaire QLQ-C30 and its lung cancer module LC-13
* To assess activity of daily life (iADL) in relation to ECOG performance status prior to study treatment
* To assess patient's outcome and treatment delivery in relation to the Charlson comorbidity score and the Simplified Comorbidity Score

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIb and IV NSCLC, excluded squamous cell NSCLC
* Age ≥ 65 years
* ECOG 0-2

Exclusion Criteria:

* Mixed, non-small cell and small cell tumours or mixed adenosquamous carcinomas with a predominant squamous component
* History of haemoptysis
* Evidence of tumour invading major blood vessels on imaging
* Radiotherapy within 28 days prior to enrolment
* Patients who are unable to interrupt aspirin or other nonsteroidal anti-inflammatory agents, other than an aspirin dose ≤ 1.3 grams per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam)
* Current or recent (within 10 days of first dose of bevacizumab) use of full-dose oral or parenteral anticoagulants or thrombolytic agent for therapeutic purposes. Prophylactic use of anticoagulants is allowed
* Clinically significant (i.e. active) cardiovascular disease for example CVA (≤6 months before enrolment), myocardial infarction (≤6 months before enrolment), unstable angina, CHF NYHA Class ≥II, serious cardiac arrhythmia requiring medication during the study and might interfere with regularity of the study treatment, or not controlled by medication
* Non-healing wound, active peptic ulcer or bone fracture
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of enrolment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 271 (Actual)
Dates: Start 2009-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Schuette, PhD MD., Study Chair — Krankenhaus Martha-Maria Halle-Doelau
Locations (1):
- Krankenhaus Martha-Maria Halle-Doelau, Halle, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab + Pemetrexed | Bevacizumab + Pemetrexed + Carboplatin
Started | 135 | 136
Completed | 92 | 98
Not Completed | 43 | 38
Not completed — Adverse Event | 17 | 22
Not completed — Death | 7 | 9
Not completed — Lack of Efficacy | 5 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — screening failure, unknown | 11 | 4

BASELINE CHARACTERISTICS:
Population: 271 patients were enrolled and randomized, due to Screening failure and subject withdrawn consent the intent-to-treat (ITT) population comprised 253 evaluable patients (BP n=119; BPC n=134).
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Pemetrexed | Bevacizumab + Pemetrexed + Carboplatin | Total
Number analyzed (Participants) | 119 | 134 | 253
Age, Continuous [Median (Full Range); unit: years] | 71.0 [65 to 86] | 72.0 [65 to 86] | 71.5 [65 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 48 | 93
  Male | 74 | 86 | 160

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival (defined as the number of days from the day of the first treatment until day of death (from any cause) or progression, whichever occurs earlier, or until the day of the last response assessment, if no progression or death (from any cause) is observed during the study).
Time Frame: 42 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Pemetrexed | Bevacizumab + Pemetrexed + Carboplatin
Number analyzed (Participants) | 119 | 134
months | 4.8 [4.3 to 6.0] | 6.8 [5.8 to 7.4]
Statistical Analysis 1: Comparison: Bevacizumab + Pemetrexed vs Bevacizumab + Pemetrexed + Carboplatin; Test type: Non-Inferiority or Equivalence — The estimation was that in the pemetrexed-carboplatin plus bevacizumab Arm the median PFS will be 5.5 months. A median PFS of 4 months (5.5 - 27%) had been regarded non-inferior. Assuming the accrual period of 24 months and the whole study duration of 42 months, 246 patients had to be recruited. According to the fact, that the required statistical power of 80% will be reached by occurrence of altogether 227 events, the final analysis was done at this time point; p = 0.0583, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 1.290, 95% CI 2-sided [0.989 to 1.682]

2. Secondary Outcome: Overall Survival
Description: Overall survival (defined as the number of days from the day of first treatment to death (from any cause), or until the last day if we know that the patient is alive).
Time Frame: 42 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Pemetrexed | Bevacizumab + Pemetrexed + Carboplatin
Number analyzed (Participants) | 119 | 134
months | 11.6 [8.6 to 14.4] | 14.4 [11.7 to 16.9]
Statistical Analysis 1: Comparison: Bevacizumab + Pemetrexed vs Bevacizumab + Pemetrexed + Carboplatin; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.3869, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 1.091, 95% CI 2-sided [0.794 to 1.499]

ADVERSE EVENTS:
Arm/Group | Bevacizumab + Pemetrexed | Bevacizumab + Pemetrexed + Carboplatin
Serious Adverse Events (participants affected / at risk) | 8/119 | 7/134
Other Adverse Events (participants affected / at risk) | 61/119 | 97/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + Pemetrexed (N=119) | Bevacizumab + Pemetrexed + Carboplatin (N=134)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 7 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + Pemetrexed (N=119) | Bevacizumab + Pemetrexed + Carboplatin (N=134)
anaemia (Blood and lymphatic system disorders) | 61 (83) | 97 (146)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No